CLINICAL TRIAL: NCT04022096
Title: A Phase 3, Double-blind, Randomized, Active-controlled Study to Evaluate the Safety and Efficacy of Tegoprazan as Maintenance Therapy in Patients With Healed Erosive Esophagitis
Brief Title: Study to Confirm the Safety and Efficacy of Tegoprazan in Patients With Healed Erosive Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJ_APA_305
Record Dates: First submitted 2019-07-14; First posted 2019-07-16 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Healed Erosive Esophagitis
MeSH Terms: interventions — tegoprazan; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tegoprazan 25mg QD (Experimental): Tegoprazan 25mg tablet, once daily, oral administration
  Interventions: Drug: Tegoprazan 25mg QD
- Lansoprazole 15mg QD (Active Comparator): Lansoprazole 15mg capsule, once daily, oral administration
  Interventions: Drug: Lansoprazole 15mg QD

INTERVENTIONS:
Drug: Tegoprazan 25mg QD — Tegoprazan 25mg tablets will be orally administered, once daily, for up to 6 months.
  Arms: Tegoprazan 25mg QD
Drug: Lansoprazole 15mg QD — Lansoprazole 15mg capsules will be orally administered, once daily, for up to 6 months.
  Arms: Lansoprazole 15mg QD

SUMMARY:
This study is designed to confirm the non-inferiority of Tegoprazan 25mg, compared to Lansoprazole 15mg as maintenance therapy in patients with healed erosive esophagitis confirmed by endoscopy following oral administration once daily(QD) for 6 months.

DETAILED DESCRIPTION:
This is a double blind, randomized, active-controlled, phase 3 study. Subjects will be randomly assigned to one of the two treatment groups (tegoprazan 25mg, lansoprazole 15mg).

ELIGIBILITY:
Inclusion Criteria:

1. Erosive eshophagitis(LA classification Grades A to D) within 12 weeks prior to Randomization
2. Healed erosive esophagitis within 7 days prior to Randomization
3. No heartburn and regurgitation within 7 days prior to Randomization

Exclusion Criteria:

1. Unable to undergo upper GI endoscopy
2. Presence of esophageal stricture, ulcerated stricture, gastroesophageal varix, long segment Barrett's esophagus with >3 cm length(LSBE), active digestive ulcer, gastric bleeding or malignant tumors on an upper GI endoscopy
3. Diagnosed with primary esophageal motility disorder, irritable bowel syndome(IBS) or inflammatory bowel disease(IBD)
4. History of acid-suppressive, esophageal or gastric surgeries

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Endoscopic remission rate of EE at 24-week | 24-week
  Endoscopic remission: No endoscopic recurrence of erosion(LA grade A to D) during maintenance period(24 weeks)

SECONDARY OUTCOMES:
Endoscopic remission rate of EE at 12-week | 12-week
  Endoscopic remission: No endoscopic recurrence of erosion(LA grades A to D) during maintenance period(12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Oh Young Lee, Ph.D, Principal Investigator — Hanyang University Seoul Hospital
Locations (1):
- Hanyang University Seoul Hospital, Seoul, South Korea